

## UNIVERSITY OF CALIFORNIA, SAN FRANCISCO SAN FRANCISCO GENERAL HOSPITAL

#### **CONSENT TO PARTICIPATE IN A RESEARCH STUDY**

## EMRLHD (Effect of Methamphetamine on Residual Latent HIV Disease) Study

This is a medical research study sponsored by the National Institutes of Health (National Institute on Drug Abuse). Your study doctor, Dr. Sulggi Lee, MD, or a member of her research team will explain this study to you.

Medical research studies include only people who choose to take part. You should take your time to make your decision about participating. You may discuss your decision with your family and friends and with your health care team. If you have any questions, you may ask your study doctor.

## You are being asked to take part in this study because:

- you have HIV infection
- you are ≥ 18 years and ≤ 65 years of age
- you are currently and have been taking antiretroviral therapy (ARVs) that include at least 3 drugs for at least the last 12 months (with no ARV changes in the last 12 weeks)
- you have had an undetectable HIV viral load for at least 12 months
- you will **not** be modifying your ARVs during the study period (146 days, approximately 5 months)
- you and your partner(s) are willing to use two forms of contraception throughout the study period as well as up to 60 days after the last day of study completion
- vou do **not** have a current or past history of methamphetamine use disorder that could put you at risk of potential return to use by participating in this study
- you are available to participate in the full study which includes 2 study treatment phases, spaced approximately 1 month apart for a total of about 146 days (approximately 5 months)
- you are **not** currently using methamphetamine or any prescription medications containing amphetamine-type stimulants (e.g., Adderall®, Dexedrine®, Ritalin®, etc.) within the last 1 year
- you do **not** have an allergy or sensitivity to amphetamine-like stimulants
- you have **not** used any other "psychoactive" drugs (cocaine, ecstasy, LSD, mushrooms, or other recreational drugs) in the last 1 month, but nicotine/tobacco, cannabis/marijuana or caffeine do not count
- you have **not** used any illicit opioids such as heroin or fentanyl in the past 3 months but prescription opioid treatments with known prescribed doses such as methadone, hydrocodone (Norco®), buprenorphine/naloxone (Suboxone®), oxycodone (Oxycontin®), or hydromorphone (Dilaudid®) are ok
- you have not recently used in the last month any medications that could potentially have a drug interaction with oral methamphetamine (e.g., an anti-depressant called a monoamine oxidase inhibitor)
- you have not had a recent hospitalization or serious infection requiring intravenous antibiotics in the last 90 days
- you are not anemic (HIV+ males Hct < 34; females Hct < 32) or contraindication to donating blood.</li>
- you do not a screening hemoglobin below 12.5 g/dL
- you do not have a history of poorly controlled high blood pressure or a systolic blood pressure >140 (after repeat measurement) in the last 3 months
- you do **not** have significant myocardial disease (e.g., current myocarditis or reduced left ventricular

ejection fraction below the lower limit of normal) or diagnose coronary artery disease.

- you do not have a prior history of heart attack or heart disease
- · you do not have an abnormal heart rhythm that needs to be medically treated
- you do **not** have a history of psychosis (e.g., hallucinations –seeing or hearing things that are not there) in the past 3 months
- you do **not** have a history of seizures, brain damage, or abnormal brain electrical activity (on electroencephalogram) in the past 3 months or currently taking anti-seizure medications
- you do not have significant history of respiratory disease requiring oxygen
- you do not have a recent history of receiving any drugs that modify the immune system in the 12 weeks prior to study
- you are **not** pregnant
- you have not had a recent vaccination within the last 2 weeks

## Why is this study being done?

This is a medical research study where we will be giving oral methamphetamine (Desoxyn®) to study participants for a single day, split into two doses. The total dose that you will receive in that single day is no more than the FDA allows children to take for the treatment of obesity.

This study is being done in HIV-infected individuals who have excellent control of their HIV in order to see if oral methamphetamine temporarily increases low levels of HIV RNA and levels of "activated" immune cells. Findings from this study may help identify ways to force persistent virus out of the body in order to achieve an HIV cure and reduce potential negative immune effects in HIV+ patients who use methamphetamine.

#### What will happen if I am in the study?

If you are in the study you will be given only one day of study medication. You will also be given one day of "placebo," or a pill that looks like the study medication but contains no active substance. After each treatment day (study medication or placebo) you will be followed for up to 31 days to study your body's response to the pill. In addition, the two treatment phases will be separated by 31 days to ensure that there is enough time for your body to "wash out" study medication (or placebo) and compare to the other treatment.

The timing of when you will receive the study medication or placebo will be randomly determined, like the toss of a coin. You will not know whether you are randomly assigned to receive the study medication first or second.

This is an open-label study, so even though you will not know when you will receive the study medication, you will know what dose of the study medication you are given. You will receive 10 milligrams of the study medication, followed by 15 milligrams of the study medication given 2 hours later, for a total dose of 25 milligrams of the study medication on the treatment day.

We will be monitoring any side effects to be sure that any side effects experienced during the study period is due to the study drug and not to other causes. In addition, based on what we know about potential drug-drug interactions between the study medication and HIV medications or other medications, you can only continue taking medically necessary medications that can be monitored during the study period. If you feel you cannot do this then you cannot enroll in this study.

# Who is paying for this study?

This study is sponsored by the National Institutes of Health (National Institute on Drug Abuse). The company that makes the study medication for this study is not involved in this research.

## How many people will take part in this study?

The study is being done in San Francisco, California. A total of 10 adults who are living with HIV will be enrolled in this study at UCSF.

## Where will I be seen for this study?

All study visits will take place at the Positive Health Program HIV/AIDS Clinic, Building 80, Wards 84/86, 995 Potrero Avenue, San Francisco or at the CTSI Clinical Research Center, Ward 5B, 1001 Potrero Avenue, San Francisco. Both clinics are at San Francisco General Hospital.

## How long will I be in this study?

The whole study will last up to 146 days. Treatment phase 1 will include one dosing day (when you receive study medication or placebo), plus 31 days of follow up. Treatment phase 1 will be followed by a 31-day "washout" period to make sure that the effects of treatment 1 is no longer in your body by the time you receive Treat 2. The washout period is also to ensure that you do not become anemic from too many blood draws during the entire 146 days of the study. Then you will receive treatment phase 2, which includes one dosing day (when you receive placebo or study medication, the opposite of what you received during treatment phase 1), plus 31 days of follow up. Your final visit will be 132 days after the first dose.



## What are my responsibilities?

Your participation in the full 146 days (approximately 5 months) of the study is critical to understand the effect of the study medication. It is very important during the entire study that you remain fully adherent to your HIV medications and do not use illicit substances or medications that would exclude you from participating in the remainder of the study. This is the reason that we perform a second screening visit at the beginning of Treatment phase 2. If you anticipate scheduling conflicts or problems in attending visits, you should notify the study doctor.

# **Detailed Summary of Study Visits:**

| screen | TREATMENT PHASE 1 | | | | | | | | washout | TREATMENT PHASE 2 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day -14 | Day -7 | Day 1 | Day 1 | Day 1 | Day 1 | Day 1 | Day 2 | Day 31 | period | Day 63 | Day 77 | Day 77 | Day 77 | Day 77 | Day 77 | Day 78 | Day 107 |
| Screen | Baseline 1 | 0 hrs | 0.5 hrs | 2 hrs | 2.5 hrs | 4 hrs | Post-24hr | Post-31d | 31 days | Baseline 2 | 0 hrs | 0.5 hrs | 2 hrs | 2.5 hrs | 4 hrs | Post-24hr | Post-31d |

## Screening Visit (Day -14)

If you agree to participate in this study you will be asked to have a screening examination at the research clinic. The screening will take approximately 1.5 hours. During the screening visit:

- You will have a complete physical examination, which will be conducted by one of the study medical staff
  to determine your health status.
- Your medical history will be documented.
- You will be asked to complete applicable HIV-related questionnaires that will ask for questions about your current and previous health, illnesses, HIV-treatment, medications, and lifestyle.
- You will also be asked to provide blood samples to check your health. Included will be tests for CD4 T-cell
  count, HIV viral load, blood count including hemoglobin, hepatitis B and C antibody, tuberculosis
  exposure, and liver, thyroid, and kidney functions.
- You will also beasked to provide a urine sample to check to be sure that you are still eligible for this study
  and have not recently used any of the substances that would exclude you from participating in the study.
- If you are a woman and you are capable of having children, a serum pregnancy testwill be performed. If this test is positive, you will not be allowed to enter the study since body changes occurring during pregnancy will alter the study results. You also agree to use a double-barrier method of contraception throughout the study period.
- You will be asked a series of extensive questions regarding any current symptoms.

The results of the screening evaluation will be reviewed to determine if you are eligible to participate in the study and you and your primary care provider will be notified of all your screening bloods results. Given the potential for changes in some of the laboratory measurements based on what time of day that you blood is drawn, it is critical that this blood draw will occur between 7:30 to 9:30 am.

#### Baseline Visit #1 (Day -7)

If you are eligible, you will return for a baseline visit. The same questionnaires that you completed at the Screening Visit will be repeated. Blood will be drawn and stored at this visit. Given the potential for changes in some of the laboratory measurements based on what time of day that you blood is drawn, it is critical that this blood draw will occur between 7:30 to 9:30 am. In addition, if you agree to provide an optional hair sample and have at least 1 inch of hair, a small thatch of hair (~300 fibers of hair) at the back of your head will be cut close to the scalp to measure the amount of HIV medications that you have been taking for approximately the last 90 days. We will also use thehair to measure for any potential substances that might exclude you from participating in the study. As at the screening visit, urine will also be collected to similarly ensure that you have not had any recent use of the substances that might exclude from participating in the study.

#### **Treatment Phase #1 Day 1 Visit**

Following randomization the first dose (the study medication or placebo) will be given on Day 1. Because the effect of the study medication on your virus is expected to be rapid and transient, you will be seen several times during the day on the Day 1 Visit. Given the potential for changes in some of the laboratory measurements based on what time of day that you blood is drawn, it is critical that this first blood draw on the treatment day occurs between 7:30 to 9:30 am. A urine sample will again be collected to ensure that you are still eligible for this study and have not recently used any of the substances that would exclude you from participating in the study.

You will have a brief physical examination and will be asked whether there has been any change in your health (illness or health problems) and whether you have taken any new medications since your last visit. In addition, an electrocardiogram (ECG) will be performed to evaluate for any abnormal electrical activity in your heart. This will occur at 0, 2, and 4 hours after you take the initial pill. You will be asked to complete a shortened version of the questionnaires you completed previously. A blood draw will be completed before the first dose is given. This blood will be used to monitor general health screening tests. A urine sample will again be collected to ensure that you are still eligible forthis study and have not recently used any of the substances that would exclude you from participating in the study. Blood will also be used to determine the amount of HIV in your blood (viral load) and the amount of white blood cells that fight infection (CD4 count). Blood will also be collected for study-specific tests including tests to measure theamount of HIV that remains in your body (even while taking HIV medications every day) and levels of inflammation in your body that might be caused by HIV.

After the seblood tests are obtained, you will be asked to take the study medication with a glass of water. For the study medication phase of the study, you will first receive 10 mg of the study medication at "hour 0" at the time of your first blood draw. You will then receive your second dose of the study medication (15 mg) at "hour 2." Your blood will be drawn at 5 timepoints on this day: 0, 0.5, 2, 2.5, and 4 hours after you take the initial pill. These frequent tests are being done as it is expected that the study medication's effect may be rapid and transient. You will be asked to stay at the study clinic for the entire visit and will be done with the treatment day approximately

1 hour after the last blood draw. The study medication will be measured in both blood and urine.

#### **Treatment Phase #1 Day 2 Visit**

You will return to the clinic for the Day 2 Visit. Given the potential for changes in some of the laboratory measurements by the time of day at which blood is drawn, it is critical that this blood draw will occur between 7:30 to 9:30 am. At this visit, you will have a single timepoint blood collection complete to monitor routine laboratory tests and to determine how much virus is in your body. A urine sample will be collected at this visit to measure methamphetamine levels after being administered the study medication (or placebo) dose the day prior. You will also have a brief physical exam, collection of vitals, health and medication questions, and completion of follow-up questionnaires.

## **Treatment Phase #1 Day 31 Visit**

You will return to the clinic 31 days from the first day of the treatment cycle. No Study medication will be given on this day. You will have a brief physical examination, will be asked if there has been any change in your health (illness or health problems), if you have missed any of your antiretroviral medications, and whether you have taken any new medications since your last visit. You will again complete the shortened version of the questionnaires you completed previously. You will have a single timepoint blood collection completed to monitor routine laboratory tests and to determine how much virus is in your body. Given the potential for changes in some of the laboratory measurements by the time of day at which blood is drawn, it is critical that this blood draw will occur between 7:30 to 9:30 am. A urine sample will again be collected to ensure that you are still eligible for this study and have not recently used any of the substances that would exclude you from participating in the study.

#### Washout Period (Day 32-62)

The washout is a 31-day period in which any effects from the first phase can resolve and return you to your pre-

study baseline state. No study procedures are completed during this period, but it is important that you continue to follow and maintain the list of inclusion criteria shown on page 1 in order to remain eligible for the remainder of the study.

## Baseline Visit #2 (Day 63)

The same procedures completed on the Day -14 Screening Visit prior to the first phase (described earlier) will be completed in preparation for the second phase.

## <u>Treatment Phase #2 Visits: Day 77 and 24-Hour Follow-up (Day 78)</u>

The same procedures that occurred on the Day 1 Visit from Phase 1 (described earlier) will occur in Phase 2 as the Day 77 and 78 Visits, respectively.

#### **Treatment Phase #2 Day 107 Follow-up Visit**

The same procedures completed on the Day 31 Follow-up Visit from Phase 1 (described earlier) will be completed for the second phase. This is the final study visit.

### **Early Withdrawal Visit**

You may discontinue the study or be withdrawn from the study at any time if you, the study doctor, or the study sponsor feels that it is not in your best interest to continue. The following is a list of possible reasons for study treatment discontinuation:

- You choose to withdraw consent and stop study participation. This is discussed in further detail later.
- The study doctor thinks it necessary for your health or safety
- You have not followed study instructions.
- The sponsor decides to stop the study.
- If you are a female of childbearing potential and have a positive pregnancy test or start breastfeeding.

For any early withdrawal from the study, you will be asked to return to the clinic for an Early Withdrawal Visit as soon as possible. At the visit you will receive a complete physical examination, vitals will be collected, medication use will be reviewed, the follow-up questionnaires will be administered, and any changes to your health will be discussed. A blood sample will be collected for clinical laboratory tests, to check your health, and to measure the amount of HIV in your body. Blood will be used to monitor routine laboratory tests and to determine how much virus is in your body.

If you are withdrawn from treatment due to a side effect or adverse event, you will be followed and treated by the study doctor until the abnormal condition or symptom has resolved or stabilized. Except in the event of withdrawal of consent, you will be asked to complete all remaining scheduled visits and procedures.

## What will happen with your blood samples?

Blood will also be sent for routine safety monitoring at most visits. HIV "viral load" and CD4+T cell counts, liver and kidney function will be measured at many visits.

By consenting to participate in this study, you consent to the storage of some of your blood samples. As part of this study, a portion of the blood obtained at some of the study visits will be stored at the UCSF AIDS Specimen Bank and/or the ARI Clinical Laboratory of Virology. Stored specimens will be sent directly to a research laboratory and/or stored for future research studies. The specimens stored for future use will be coded. This code will be kept confidential and only Dr. Lee and her research collaborators will have access to these specimens and key linking them to the study participants.

Future studies using your specimens may be performed by scientists based at the University of California, San Francisco and/or by scientists based at other institutions, such as other universities, the NIH and commercial laboratories. All efforts to minimize personally identifying information will be carried out. No personal identifiers will be kept with your sample or shared with other researchers. The possible types of studies which may be performed include tests for infections that are common in HIV-infected patients such as cytomegalovirus or human herpesvirus 8, genetic testing, as well as new tests measure the amount of "latent" HIV reservoir (the very low amounts of virus that remain in your body despite you taking antiretroviral therapy and having "undetectable" viral loads on your clinical labs).

If you agree, any information obtained from the laboratory studies that may be important for your clinical care will be shared with you and/or your primary care provider, but research-related results that are currently unimportant to your clinical care will not be shared with you, as they are exploratory in nature. Specimens will be kept until they are used up or destroyed For the current study, the following research tests may be performed: (1) the activation level of your T cells, (2) the amount of HIV in your blood, and (3) the amount of HIV in your cells. Other tests related to this study, which are unknown at this time, may be performed. Results from the research performed on these samples for this study and/or future studies will not be shared with you, as they are experimental in nature. However, you can receive results of standard laboratory tests performed by the study, such as CD4+ T cell counts, routine HIV viral load tests, etc.

Donating data may involve a loss of privacy, but information about you will be handled as confidentially as possible. Study data will be physically and electronically secured. As with any use of electronic means to store data, there is a risk of breach of data security.

There will be no direct benefit to you from allowing your data to be kept and used for future research. However, we hope we will learn something that will contribute to the advancement of science and understanding of health and disease. If the data or any new products, tests or discoveries that result from this research have potential commercial value, you will not share in any financial benefits. If you decide later that you do not want your information to be used for future research, you can notify the investigator in writing (sulggi.lee@ucsf.edu or 995 Potrero Avenue, Building 80, Box 0874, San Francisco, CA 94110), and any remaining specimens and data will be destroyed. However, we cannot retract any data has been shared with other researchers.

### Can I stop being in the study?

Your participation in this study is voluntary. If you do participate, you may freely withdraw from the study at any time. Your decision will not change your future medical care at any of the study sites or at the San Francisco General Hospital.

Your participation in this study may be stopped at any time by the study doctor or the sponsor without your consent. The reasons might include:

- the study doctor thinks it necessary for your health or safety; you have not followed study instructions;
- the sponsor has stopped the study; or administrative reasons require your withdrawal.

If you leave the study before the final regularly scheduled visit, you may be asked by the study doctor to make a final visit for some of the end of study procedures.

IRB NUMBER: 18-26765 IRB APPROVAL DATE: 02/03/2022 ilty of California IRB EXPIRATION DATE: 02/02/2023

## What if I become pregnant during this study?

You should not become pregnant or father a baby while on this study, because the study medication may affectan unbornbaby. If you are a woman and you are capable of having children, a pregnancy test will be performed. If this test is positive, you will not be allowed to enter the study. Women should not breastfeed a baby while on this study. It is important to understand that you need to use birth control while on this study. You must agree to use at least two effective methods of contraception throughout the study period and up to 90 days after the last dose of study treatment. Since there are limited data on pregnancy risk related to methamphetamine given for a single day at the FDA-approved pediatric daily dose, we will take precautions around potential pregnancy during the trial.

If a participant is able to become pregnant, two of the following forms of birth control are required, one of which must be condoms or a diaphragm or cervical cap:

- Condoms (male of female) with or without a spermicidal agent
- Diaphragm or cervical cap with spermicide
- Intrauterine device (IUD)—this must be a brand that has a reported failure rate is < 1% per year
- Tubal ligation
- Hormone-based contraceptive such as oral birth control pills

If you are a female and become pregnant during the clinical trial, you are advised:

- To call/notify the study doctor immediately
- To consult an obstetrician or maternal-fetal specialist
- You will not be given any additional investigational products
- You will be followed to determine the pregnancy outcome

If you are a male who is sexually active with a woman capable of becoming pregnant, you must agree to use a medically accepted form of birth control during the course of this research study. You must inform your partner of the potential harm to an unborn child. Your partner needs to know that if she does become pregnant during the study:

- You will need to call/notify the study doctor immediately
- She will need to consult an obstetrician or maternal-fetal specialist
- Study staff will ask for her permission to collect information about the pregnancy and the health of the baby. This includes information related to the pregnancy/delivery and obstetrical history.

If you or your partner become pregnant while on study, you must tell the study staff right away and stop taking the study medication. You (or your partner) should also see your doctor to get the best care possible. You may remain on study during your pregnancy or you may leave the study. Either way, the study staff will contact you to find out about any events that happen during the pregnancy and about the health of the baby.

#### What side effects or risks can I expect from being in the study?

If you decide to participate in this study, you will receive the study medication for 1 day. You will be required to remain on your stable antiretroviral regimen throughout the study. Below is a description of most of the side effects that may occur during this study, but not all possible side effects.

What are potential risks and discomforts from participating in the study?

Side effects associated with taking the study medication

Likely to occur:



IRB NUMBER: 18-26765 IRB APPROVAL DATE: 02/03/2022 University of California IRB EXPIRATION DATE: 02/02/2023
San Francisco

Oral methamphetamine is a stimulant and may cause increased blood pressure, heart rate, and palpitations (noticeably rapid, strong, or irregular heartbeats). Less likely to occur:

 In some cases, oral methamphetamine can cause some dizziness, headache, insomnia, elevated mood, depressed mood, restlessness, diarrhea, constipation, unpleasant taste, dry mouth, and tremor (hands shaking).

## Very unlikely to occur:

- At very high doses (much higher than the doses being given in this study) and if taken for
  prolonged periods of time (e.g., weeks to months to years), oral methamphetamine can lead
  to a substance use disorder, exacerbation of preexisting abnormal movements (called "tics"),
  psychotic symptoms (hearing and seeing things that are not actually there), frequent
  erections, impotence, and changes in libido.
- Long-term effects that cannot be known

# $Side effects\,associated\,with\,taking\,Place bo$

Very unlikely tooccur:

In order to make the placebo appear similar to the study medication, the pills will be crushed
and placed in a capsule. For the placebo phase, cornstarch will be placed inside the capsule.
Therefore, individuals who have an allergy to cornstarch may be at risk of an allergic reaction
when taking placebo and should notify the study investigator if they have a known allergy to
corn starch.

Wewill be monitoring your response to the study drug very closely. In the event of a serious adverse event, we will provide you appropriate medical care immediately.

## HIV viral load and resistance to antiretroviral therapy risks

• We will be measuring the amount of viral RNA that increases in your blood after giving you the study drug. This does not necessarily mean that there is an increase in the amount of circulating HIV. Nonetheless, since there is a very small chance that the study drug might transiently increase you HIV viral load, there would be a theoretical risk of developing resistance to antiretroviral therapy and of transmitting HIV to uninfected persons if you were not on a stable regimen and adequately suppressed on your ARVs. The likelihood of this is extremely low, given that you will only be given one day of a single day's maximum (child) dose of the study medication, and if the study medication causes your viral load to increase, the predicted increases in HIV in the blood is extremely small. For these reasons, you can only participate in this study if there are alternate ART regimens available in the rare event that your current ART regimen is compromised as a result of this study. During the study, you will also have your HIV viral load followed closely (at screening, baseline, and on days 2, and 31 of each treatment arm).

#### Drug-drug interactions

• The following medications are not allowed during the study because of potential interactions with the study medication: acebrophyline, iobenguane, isocarboxazid, methylene blue, moclobemide, phenylzine, procarbazine, rasagiline, safinamide, selegiline, tranylcypromine, asunaprevir, buproprion, topical cocaine, fluoxetine, iohexol, linezolid, paroxetine, potassium citrate, quinidine, sodium bicarbonate, sodium citrate, sodium lacate, tipranavir, and tromethamine. This is because the study medication may alter metabolism of the drugs.

## Side effects of taking your blood sample (phlebotomy)

Likely to occur:

Drawing blood from a vein may cause some discomfort, bleeding or bruising where the needle

enters the skin, and rarely, fainting or infection may occur. Up to a total of 795 milliliters (about 53 tablespoons) will be collected during the course of this study, and the maximum volume of blood per visit will be 52 milliliters, all of which has been carefully calculated over the 146 days of the study to ensure that your blood levels are not below American Red Cross Guidelines.

### Less likely to occur:

Less common symptoms include lightheadedness, dizziness, fainting and nausea. Symptoms of anemia include tiredness, weakness and dizziness. You will be checked for anemia at all visits from screening through day 31 of each treatment arm. If the investigator feels that you are at significant risk for anemia, the amount of blood collected will be reduced. If your hemoglobin falls below 10 g/dl or your hematocrit falls below 27%, you will have 5 ml (1 teaspoon) of blood drawn to check your hemoglobin and hematocrit. Other than the blood required to check your hemoglobin and hematocrit, you will not have more blood drawn until your hemoglobin rises above 10 g/dl or your hematocrit rises above 27%

We will measure your baseline hemoglobin to ensure that it is safe for you to participate in this study. In order to participate in this study, your baseline hemoglobin must be >12 g/dl. You should know that the prediction of side effects in any individual cannot be done with certainty and unexpected potentially harmful effects occasionally occur with the administration of any type of drug or study procedure. If serious side effects occur, the study will be stopped.

#### Confidentiality

Participation in research may involve a loss of privacy; however, your records will be handled as confidentially as possible. All study questionnaires and research samples will be coded with a study ID. No personal identifiers such as your name will be used for stored specimens. Dr. Lee and the research staff as well as the UCSF Institutional Review Board will have access to your study records and test results. In addition, your records may be inspected by the Research Advisory Panel of California. No individual identities will be used in any reports or publications that may result from this study. California regulations require laboratories to report new cases of tuberculosis, hepatitis B, and hepatitis C infection to the county public health department. The reports include the patient's name, social security number, and other identifying information. Information about these new infections is used to track these diseases statewide and nationwide. Other than this required reporting, your results will be treated confidentially by the study staff. Personally identifying information will not be reported to other departments or agencies.

#### Are there benefits to taking part in the study?

This study will not provide you with any direct benefit. It is hoped that this study will help learn how to reduce the total amount of HIV in the body, but this may not happen. This study will not result in a cure.

#### What other choices do I have if I do not take part in this study?

The alternative to this study is to choose not to participate.

#### Will my medical information be kept private?

Records of this study will be kept confidential and you will not be identified in any written or verbal reports with the following possible exceptions. Your records may be inspected by the UCSF Institutional Review Board (IRB), which is a committee that watches over the safety and rights of research subjects or the Food and Drug Administration (FDA) if required for an internal audit, National Institute of Health (NIH), Office of Human Research Protections (OHRP). Your confidentiality will be protected in accordance with applicable research practice. All research records will be kept in locked files located within locked rooms to which only study staff have

access and/or within limited access, computer files available only to investigators and study personnel. Your name will be removed from all research study records. Only initials and code numbers will be present on study records and documents. Any publication or presentation of study results will not identify you by name. A medical record is created when you are admitted to the Clinical Research Center at San Francisco General Hospital. This record will have personally identifying information in it, but will be kept confidential, as would any hospital medical record.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Participation in research can cause a loss of privacy. In this study you will be asked about drug use and other possibly illegal activities. The researcher will keep information about you as confidential as possible, but complete confidentiality cannot be guaranteed. On rare occasions, research records have been subpoenaed by a court.

## What are the costs of taking part in this study?

There are no charges for the study visits. Any laboratory tests and visits required by the study will be provided at no cost to you. You will receive the study drug free of charge. Neither you nor your insurance company will be responsible for any study-associated costs.

#### Will I be paid for taking part in this study?

Yes. You will be paid for each visit. If you are eligible for this study and choose to participate, in return for your time, effort, and travel expenses, you will be paid \$35 in cash or with amazon e-code at the completion of each standard study visit. If you agree to the optional hair collection, you will be paid \$25 in cash or amazon e-code for a small sample of hair collected at the baseline 1 and 2 visits only. Due to the length of time required for the study medication (and placebo) dosing days, for these visits you will be paid \$150 (as amazon e-code or as \$50 in cash and \$100 by check) at the completion of each (the study medication or placebo administration phase) day and also be provided with a meal and refreshments. This is a total of up to \$630 for completion of all study visits. We will need your social security number to report the income to the Internal Revenue Services if the total amount of research compensation for the study exceeds \$600 in one calendar year.

## What happens if I am injured because I took part in this study?

It is important that you tell the study doctor, Dr. Sulggi Lee, if you feel that you have been injured because of taking part in this study. You can tell the doctor in person or call her at (415) 735-5127.

**Treatment and Compensation for Injury:** If you are injured as a result of being in this study, the University of California will provide necessary medical treatment. The costs of the treatment may be billed to you or your insurer just like any other medical costs, or covered by the University of California, depending on an umber of factors. The University does not normally provide any other form of compensation for injury. For further information about this, you may call the UCSF Institutional Review Board at 415-476-1814.

#### What are my rights if I take part in this study?

Taking part in this study is your choice. You may choose either to take part or not to take part in the study. If you decide to take part in this study, you may leave the study at any time. No

HIV methamphetamine study

Prepared 06/20/2021



matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits. Leaving the study will not affect your medical care. You can still receive your medical care from our institution.

We will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

In the case of injury resulting from this study, you do not lose any of your legal rights to seek payment by signing this form.

# Who can answer my questions about the study?

In the future, you may have questions about your study participation. You may also have questions about a possible side effect, reaction to study medication, or a possible research-related injury. If you have any questions, please contact Dr. Lee (the study investigator) at phone: (415) 735-5127, email: <a href="mailto:sulggi.lee@ucsf.edu">sulggi.lee@ucsf.edu</a>

For questions about your rights while taking part in this study, you can call the UCSF Institutional Review Board (a group of people who review the research to protect your rights) can be reached at (415) 476-1814.

Do not sign this consent form unless you have had a chance to ask questions and have received satisfactory answers to all of your questions.



#### CONSENT

You have been given copies of this consent form and the Experimental Subject's Bill of Rights to keep. PARTICIPATION IN RESEARCH IS VOLUNTARY. You have the right to decline to participate or to withdraw at any point in this study without penalty or loss of benefits to which you are otherwise entitled.

You will be asked to sign a separate form authorizing access, use, creation, or disclosure of health information about you. I have read this information, which is printed in English. This is a language that I read and understand. Participant Name, printed Participant Signature Date SignatureofPersonConductingInformedConsentDiscussion Date **CONSENT FOR GENETIC TESTING** Genetic information (also known as genotype data) and the medical record data (also known as phenotype data) may be shared broadly in a coded form for future genetic research or analysis. We may give certain medical information about you (for example, diagnosis, blood pressure, age if less than 85) to other scientists or companies not at UCSF, including to a public government health research database, but we will not give them your name, address, phone number, or any otheridentifiable information. Research results from these studies will not be returned to you, as they are exploratory in nature. Results of this testing will not be available to you or your providers, just to the researchers in the study. Genetic information that results from this study does not have medical or treatment importance at this time. However, there is a risk that information about taking part in a genetic study may influence insurance companies and/or employers regarding your health. Taking part in a genetic study may also have a negative impact or unintended consequences on family or other relationships. It is possible that future research could one day help people of the same race, ethnicity, or sex as you. However, it is also possible through these kinds of studies that genetic traits might come to be associated with your group. In some cases, this could reinforce harmful stereotypes. Please indicate below if you do not agree to genetic testing on the sample collected for this study. (initials) YES, lagree (initials) NO, I do not agree

# CONSENT FOR HAIR SAMPLE COLLECTION

Drug levels in hair samples can tell research investigators how much medication gets into a person's body. For this study, you will be asked to have a small sample of hair (about 200 strands)



IRB NUMBER: 18-26765 IRB APPROVAL DATE: 02/03/2022 rsity of California IRB EXPIRATION DATE: 02/02/2023

cut from your head so that we can measure levels of HIV drugs in this small hair sample. Levels in hair may give us a better idea of long-term exposure to a drug. Of note, humans lose about 100 hairs from their head every day naturally so this amount of hair removal should not be noticeable. There is a small chance of cutting or nicking the scalp from the cutting of the hair sample. This process will not be disruptive to your hairstyle. Results of this testing will not be available to you or your providers, just to the researchers in the study.

| Please indica study. | ate below if you do not ag | greetohavea | small amount of your hair collected for this |
|---|---|---|---|
| (ini | tials)YES,Iagree | | _(initials) NO, I do not agree |
| Drug levels ir<br>person's bod<br>at each study<br>marijuana, ar | y over the past few days<br>visit so that we can mea | research inve<br>s. For this stud<br>sure levels of | estigators how much medication gets into a<br>ly, you will be asked to provide a urine sample<br>drugs, including methamphetamine, cocaine,<br>not be available to you or your providers, just to |
| Please indic | ate below if you do not | t agree to ha | ve urine collected for this study. |
| (ini | tials)YES,Iagree | | _(initials) NO, I do not agree |



The rights below are the rights of every person who is asked to be in a research study. As an experimental subject I have the following rights:

- 1) To be told what the study is trying to find out,
- 2) To be told what will happen to me and whether any of the procedures, drugs, or devices is different from what would be used in standard practice,
- 3) To be told about the frequent and/or important risks, side effects, or discomforts of the things that will happen to me for research purposes,
- 4) To be told if I can expect any benefit from participating, and, if so, what the benefit might be,
- 5) To be told of the other choices I have and how they may be better or worse than being in the study,
- 6) To be allowed to ask any questions concerning the study both before agreeing to be involved and during the course of the study,
- 7) To be told what sort of medical treatment is available if any complications arise,
- 8) To refuse to participate at all or to change my mind about participation after the study is started. This decision will not affect my right to receive the care I would receive if I were not in the study,
- 9) To receive a copy of the signed and dated consent form,
- 10) To be free of pressure when considering whether I wish to agree to be in the study.

If I have other questions I should ask the researcher or the research assistant. In addition, I may contact the Institutional Review Board, which is concerned with protection of volunteers in research projects. I may reach the committee office by calling: (415) 476-1814 from 8:00 AM to 5:00 PM, Monday to Friday, or by writing to the UCSF Human Research Protection Program, Box 0962, 3333 California St., Ste. 315, San Francisco, CA 94143.

Call 476-1814 for information on translations.